CLINICAL TRIAL: NCT01102972
Title: A Prospective, Randomized, Multicenter, Open-Label Study to Compare the Efficacy and Safety of Simplifying From a Regimen of Atazanavir (ATV) + Ritonavir (RTV) + Tenofovir/Emtricitabine to ATV + Abacavir/Lamivudine Without RTV in Virologically Suppressed, HIV-1 Infected, HLA-B*5701 Negative Subjects
Brief Title: A Simplification Study of Unboosted Reyataz With Epzicom (ASSURE)
Acronym: ASSURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113734
Record Dates: First submitted 2010-04-08; First posted 2010-04-13 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-09

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: HIV-1; HIV
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — Atazanavir Sulfate; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATV + ABC/3TC (Experimental): Subjects will change to ATV 400mg administered as two 200mg capsules orally, once daily and to the fixed-dose combination tablet of ABC 600mg/3TC 300mg (EPZICOM) administered as one tablet orally, once daily for 48 weeks. The subject's pre-study RTV will be discontinued.
  Interventions: Drug: Reyataz + Epzicom
- ATV + RTV + TDF/FTC (Active Comparator): Subjects will continue their pre-study therapy, un-modified, of ATV 300mg administered as one capsule orally, once daily plus RTV 100mg administered orally, once daily plus fixed dose combination tablet tenofovir 300mg/emtricitabine 200mg administered as one tablet orally, once daily for 48 weeks.
  Interventions: Drug: Reyataz + Norvir + Truvada

INTERVENTIONS:
Drug: Reyataz + Norvir + Truvada — atazanavir 300mg + ritonavir 100mg + tenofovir 300mg/emtricitabine 200mg
  Arms: ATV + RTV + TDF/FTC
Drug: Reyataz + Epzicom — atazanavir 400mg + abacavir 600mg/lamivudine 300mg
  Arms: ATV + ABC/3TC

SUMMARY:
This study is designed to compare the efficacy and safety of simplifying therapy from a regimen of atazanavir (ATV) + ritonavir (RTV) + tenofovir/emtricitabine (TDF/FTC) to a regimen of ATV + abacavir sulfate/lamivudine (ABC/3TC) without RTV in virologically suppressed, HIV-1 infected, HLA-B*5701 negative subjects for 48 weeks.

DETAILED DESCRIPTION:
A prospective, randomized, multicenter, open-label study to compare the efficacy and safety of simplifying from a regimen of atazanavir (ATV) + ritonavir (RTV) + tenofovir/emtricitabine (TDF/FTC) to ATV + abacavir sulfate/lamivudine (ABC/3TC) without RTV for 48 weeks in virologically suppressed, HIV-1 infected, HLA-B*5701 negative subjects.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult (greater than or equal to 18 years) with documented HIV-1 infection
* Subject is a male or female of non-childbearing potential (physiologically incapable of becoming pregnant, is pre-menarchal or post-menopausal) or child-bearing potential with a negative pregnancy test who agrees to avoid pregnancy by sexual abstinence or utilization of a highly effective method of birth control throughout the study period
* Subject is receiving a once-daily regimen of ATV (300mg) + RTV (100mg) + TDF/FTC (300mg/200mg) for at least 6 months prior to or by the first day of screening. ATV + RTV + TDF/FTC must be the subejct's INITIAL regimen or FIRST or SECOND SWITCH regimen. If ATV + RTV + TDF/FTC is subject's first or second switch regimen, then subject may ONLY have received the following prior regimens: a) any currently licensed non-nucleoside reverse transcriptase inhibitor (NNRTI) + TDF/FTC or ZDV/3TC; b) RTV-boosted PI with TDF/FTC or ZDV/3TC; or c) an alternative regimen not listed above after approval by Sponsor.
* Subject is virologically suppressed on ATV + RTV + TDF/FTC defined as HIV-1 RNA </=75 copies/mL at 2 consecutive timepoints, one of which is at Screening and the other at least 28 days prior to Screening

Exclusion Criteria:

* Subject has evidence of virologic failure
* Subject has any known HIV genotyping results indicating HIV virus contains any of the following resistance mutations in reverse transcriptase including K65R, K70E, L74V, M184I/V or Y115F, a combination of two or more thymidine analog mutations including M41L, D67N, K70R, K219Q or E that include changes at either L210 or T215), or 3 or more of the following HIV-1 protease mutations associated with atazanavir resistance: D30, V32, M36, M46, I47, G48, I50, I54, A71, G73, V77, V82, I84, N88, and L90
* Subject is HLA-B*5701 positive
* Subject has hypersensitivity to any component of the study drugs
* SUbject is pregnant or breastfeeding
* Subject is enrolled in one or more investigational drug protocols within 30 days of screening
* Subject has an active Center for Disease Control and Prevention (CDC) Category C disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy during the trial
* Subject has ongoing clinically relevant hepatitis at screening and/or positive for Hepatitis B (+ HbsAg)
* Subject has a creatinine clearance <50 mL/min via the Cockcroft-Gault method
* Subject has a verified Grade 4 laboratory abnormality at screening unless the Investigator can provide a compelling explanation (e.g. elevated CPK due to exercise) for the laboratory result(s) and has the assent of the Sponsor
* Subject has any other laboratory abnormality or medical condition at screening, which, in the opinion of the investigator, would preclude the subject's participation in the study
* Subject has had an immunization within 30 days prior to first dose of investigational product
* Subject has had any exposure to treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, or interferons) or receipt of an HIV-1 immunotherapeutic vaccine within 90 days prior to screening. Subjects using inhaled corticosteroids or short-course systemic corticosteroids (less than or equal to 14 days) are eligible for enrollment.
* Subject has had treatment with radiation therapy or cytotoxic chemotherapeutic agents within 90 days prior to screening, or has an anticipated need for these agents within the study period
* Subject has had treatment within 30 days prior to first dose of investigational product for or an anticipated need during the study of any medications which can have interactions with the study medications, TDF, FTC, ABC, 3TC, ATV and/or RTV, as described in current product labelling
* Subject has had treatment with any previous abacavir-containing regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2010-04; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (41):
- United States (39):
  - GSK Investigational Site, Hobson City, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Wilton Manors, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Berkeley, Michigan
  - GSK Investigational Site, East Lansing, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Spokane, Washington
- Puerto Rico (2):
  - GSK Investigational Site, Ponce, Puerto Rico
  - GSK Investigational Site, San Juan, Puerto Rico

REFERENCES:
- [Background] Robertson K, Maruff P, Wohl D, et al. Similar cognition outcomes after 24 weeks for tenofovir/FTC + atazanavir/r (ATV/r)-experienced HIV+ subjects or subjects simplifying to abacavir/3TC+ATV. Published at: Conference on Retroviruses and Opportunistic Infections - 20th Annual; March 3-6, 2013; Atlanta, GA.
- [Result] D. Wohl, L. Bhatti, P. Maruff, K. Robertson, C. Small, H. Edelstein, H. Zhao, D. Margolis, L. Ross, M. Shaefer, on behalf of the ASSURE (EPZ113734) Study Team. Prevalence of HIV Associated Neurocognitive Disorders (HAND) in Virologically Suppressed HIV+ Individuals. 19th International AIDS Conference; July 22-27, 2012; Washington, DC. Poster WEPE092.
- [Result] C. B. Small, D. Wohl, D. A. Margolis, B. Wine, L. L. Ross, H. Zhao, and M. S. Shaefer. Prevalence of HLA-B*5701 Allele in HIV-infected Subjects in North America and Reductions in Risk for Development of Abacavir Associated Hypersensitivity Reaction (ABC HSR). 52nd Interscience Conference on Antimicrobial Agents and Chemotherapy; September 9-12, 2012; San Francisco, CA. Poster H-895
- [Result] D. Wohl, L. Bhatti, C. B. Small, H. Edelstein, H. Zhao, D. A. Margolis, L. L. Ross, M.S. Shaefer. Simplification to Abacavir/Lamivudine (ABC/3TC) + Atazanavir (ATV) from Tenofovir/Emtricitabine (TDF/FTC) + ATV/Ritonavir (RTV, /r) Maintains Viral Suppression and Improves Bone Biomarkers. 52nd Interscience Conference on Antimicrobial Agents and Chemotherapy; September 9-12, 2012; San Francisco, CA. Oral presentation H-556c.
- [Derived] Small CB, Margolis DA, Shaefer MS, Ross LL. HLA-B*57:01 allele prevalence in HIV-infected North American subjects and the impact of allele testing on the incidence of abacavir-associated hypersensitivity reaction in HLA-B*57:01-negative subjects. BMC Infect Dis. 2017 Apr 11;17(1):256. doi: 10.1186/s12879-017-2331-y. PMID 28399804
- [Derived] Wohl DA, Bhatti L, Small CB, Edelstein H, Zhao HH, Margolis DA, DeJesus E, Weinberg WG, Ross LL, Shaefer MS. Simplification to abacavir/lamivudine + atazanavir maintains viral suppression and improves bone and renal biomarkers in ASSURE, a randomized, open label, non-inferiority trial. PLoS One. 2014 May 13;9(5):e96187. doi: 10.1371/journal.pone.0096187. eCollection 2014. PMID 24825167
- See also: ViiV Healthcare Website — http://www.viivhealthcare.com
- See also: Click here for more information about Epzicom — http://www.epzicom.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (PAR) were recruited from 44 centers in the United States, including Puerto Rico. ATV, atazanavir; RTV, ritonavir; TDF, tenofovir; FTC, emtricitrabine; QD, once daily; HIV-RNA, human immunodeficiency virus-ribonucleic acid; c, copies; ml, milliliters; ART, antiretroviral; mg, milligrams, ABC/3TC, abacavir sulfate/lamivudine.
Pre-assignment Details: HLA-B*5701-negative PAR receiving an ATV/RTV + TDF/FTC regimen QD who are virologically suppressed (plasma HIV-1 RNA <75 c/mL) and met all eligibility requirements were randomized 2:1 to receive an ART regimen of ATV 400 mg QD + ABC/3TC 600 mg/300 mg QD (simplification arm) or ATV/RTV 300 mg/100 mg QD + TDF/FTC 300 mg/200 mg QD (continuation arm).
Groups:
- ABC/3TC + ATV: Abacavir (ABC) 600 milligrams (mg)/lamivudine (3TC) 300 mg fixed-dose combination tablet (FDC) once a day (QD) plus atazanavir (ATV) 400 mg (given as oral capsules) QD for 48 weeks
- TDF/FTC + ATV/RTV: Tenofovir (TDF) 300 mg/Emtricitabine (FTC) 200 mg FDC tablet QD plus Atazanavir (ATV) 300 mg (given as oral capsules)/Ritonavir (RTV) 100 mg (given as oral capsules) QD for 48 weeks
Period: Overall Study
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Started | 199 (297 PAR enrolled. 1 PAR withdrew before taking investigational product and didn't "start" the study.) | 97 (297 PAR enrolled. 1 PAR withdrew before taking investigational product and didn't "start" the study.)
Completed Week 24 | 180 | 88
Completed | 170 (These participants completed Study Week 48.) | 83 (These participants completed Study Week 48.)
Not Completed | 29 | 14
Not completed — Adverse Event | 8 | 2
Not completed — Lack of Efficacy | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 10 | 5
Not completed — Investigator Discretion | 2 | 0
Not completed — Withdrawal by Subject | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV | Total
Number analyzed (Participants) | 199 | 97 | 296
Age Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (9.54) | 42.3 (10.20) | 42.6 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 18 | 62
  Male | 155 | 79 | 234
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 26 | 77
  Not Hispanic or Latino | 148 | 71 | 219
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 65 | 37 | 102
  American Indian or Alaskan Native | 3 | 0 | 3
  Asian - East Asian Heritage | 2 | 0 | 2
  Asian - South East Asian Heritage | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White - Arabic/North African Heritage | 2 | 0 | 2
  White - White/Caucasian/European Heritage | 120 | 55 | 175
  Mixed Race | 3 | 3 | 6
Number of participants with the indicated baseline HIV-RNA level [Number; unit: participants] — HIV-1 RNA, Human Immunodeficiency Virus type 1 Ribonucleic acid. HIV-1 viral load was measured as virus copies per milliliter (mL) at baseline.
  participants
    HIV-1 RNA <50 | 192 | 93 | 285
    HIV-1 RNA 50-<75 | 2 | 2 | 4
    HIV-1 RNA >=75 | 5 | 2 | 7
Number of participants with the indicated Baseline CD4+ Cell Count [Number; unit: participants] — A CD4+ cell is a T lymphocyte that carries the CD4 antigen. Immunologic response was assessed by CD4+ counts, measured as the number of cells per cubic millimeter.
  participants
    CD4+ cells <50 | 0 | 0 | 0
    CD4+ cells 50-<200 | 14 | 6 | 20
    CD4+ cells >=200 | 185 | 91 | 276
Number of participants with the indicated Center for Disease Control (CDC) Classification [Number; unit: participants] — Acquired Immunodeficiency Syndrome (AIDS) CDC classifications are Asymptomatic, Symptomatic, or AIDS. The CDC categorization of HIV/AIDS is based on the lowest documented CD4 cell count (Class A, >=500 cells per microliter [µl]; Class B, 200-499 cells/µl; Class C, <200 cells/µl) and on previously diagnosed HIV-related conditions.
  participants
    Class A: Asymptomatic/lymphadenopathy/acute HIV | 136 | 67 | 203
    Class B: Symptomatic, not AIDS | 26 | 13 | 39
    Class C: AIDS indicator conditions | 37 | 17 | 54
Median Baseline CD4+ Cell Count [Median (Full Range); unit: cells per cubic millimeter] | 492.0 [77.0 to 1196.0] | 480.0 [108.0 to 1479.0] | 491.5 [77.0 to 1479.0]
Median Baseline HIV-1 RNA Level [Median (Full Range); unit: log10 copies/mL] | 1.591 [1.591 to 3.900] | 1.591 [1.591 to 3.285] | 1.591 [1.591 to 3.900]
Number of participants with the indicated Baseline Hepatitis B (HB) Status [Number; unit: participants] — The HB surface antigen is a protein present on the surface of the hepatitis B virus (HBV). It can be detected in the blood of participants with acute and chronic HBV infections. A non-reactive test result likely means that participants are not infected with HB, but does not exclude the possibility of exposure to or infection with HB.
  participants
    Reactive | 0 | 0 | 0
    Non-reactive | 199 | 97 | 296
Number of participants with the indicated Baseline Hepatitis C (HC) Status [Number; unit: participants] — The HC surface antigen is a protein present on the surface of the hepatitis C virus (HCV). It can be detected in the blood of participants with acute and chronic HCV infections. A non-reactive test result likely means that participants are not infected with HC, but does not exclude the possibility of exposure to or infection with HC.
  participants
    Reactive | 18 | 8 | 26
    Non-reactive | 181 | 89 | 270

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants (PAR) Who Achieved Plasma HIV-1 RNA <50 Copies (c)/Milliliter (mL) at the Week 24 Visit: TLOVR Analysis
Description: The percentage of PAR with HIV-1 RNA virus <50 c/mL determined from blood samples drawn at Week 24 was tabulated by treatment arm with stratification by initial antiretroviral treatment. Per TLOVR algorithm, responders were PAR with confirmed viral load <50 c/mL who had not met any non-responder criterion. Non-responders were PAR who never achieved confirmed HIV RNA <50 c/mL, prematurely discontinued study or study medication for any reason, had confirmed rebound to at least 50 c/mL, or had an unconfirmed HIV RNA of at least 50 c/mL at the last visit.
Time Frame: Week 24
Population: Intent-to-Treat (ITT)-Exposed Population: all participants exposed to at least one dose of study medication. The primary analysis method was time to loss of virologic response (TLOVR) for the proportion of participants HIV-1 RNA <50 copies/mL at Week 24.
Measure: Number; unit: percentage of participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
percentage of participants | 86.9 | 86.6
Statistical Analysis 1: Comparison: ABC/3TC + ATV vs TDF/FTC + ATV/RTV; Test type: Non-Inferiority or Equivalence — Non-inferiority would be established between the two arms if the lower limit of the 2-sided 95% confidence interval (CI) for the difference in the percentage of participants with HIV-1 RNA <50 copies/mL at Week 24 was -12% or greater; p = 0.937, Cochran-Mantel-Haenszel — The p-value was obtained from the Cochran-Mantel-Haenszel method stratified by initial antiretroviral regimen; Treatment difference of proportions = 0.33, 95% CI [-7.97 to 8.64] — 95% confidence intervals were calculated (using Mantel-Haenszel weight) stratified by initial antiretroviral regimen

2. Secondary Outcome: Percentage of Participants (PAR) Who Achieved Plasma HIV-1 RNA <50 c/mL at the Week 24 Visit: Observed, M/D=F, and SNAPSHOT Analyses
Description: The percentage of PAR with HIV-1 RNA virus <50 c/mL determined from blood samples drawn through Week 24 was tabulated by treatment arm with stratification by initial antiretroviral treatment using specific analysis methods.
Time Frame: Week 24
Population: ITT-E Population. Analysis methods: (1) Observed: all observed data; (2) missing or discontinuation equals failure (M/D=F): PAR with missing data/data collected after study medication discontinuation (DC) were failures; (3) SNAPSHOT: PAR with missing data at Week 24/data collected after study medication DC/viral load >=50 c/mL were failures.
Measure: Number; unit: percentage of participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
percentage of participants
  Observed, n=181, 89 | 94.5 | 97.7
  M/D=F, n=199, 97 | 84.9 | 87.6
  SNAPSHOT, n=199, 97 | 84.9 | 88.7

3. Secondary Outcome: Percentage of Participants (PAR) Who Achieved Plasma HIV-1 RNA <50 c/mL at the Week 48 Visit: TLOVR, Observed, M/D=F, and SNAPSHOT Analyses
Description: The percentage of PAR with HIV-1 RNA virus <50 c/mL determined from blood samples drawn at Week 48 was tabulated by treatment arm with stratification by initial antiretroviral treatment using specific analysis methods.
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
Percentage of participants
  TLOVR, n=199, 97 | 76.4 | 79.4
  Observed, n=169, 82 | 91.1 | 96.3
  M/D=F, n=199, 97 | 76.9 | 79.4
  SNAPSHOT, n=199, 97 | 77.4 | 81.4

4. Secondary Outcome: Percentage of Participants (PAR) Who Achieved Plasma HIV-1 RNA <400 c/mL at the Week 24 Visit: TLOVR Analysis
Description: The percentage of PAR with HIV-1 RNA virus <400 c/mL determined from blood samples drawn at Week 24 was tabulated by treatment arm with stratification by initial antiretroviral treatment. Per TLOVR algorithm, responders were PAR with confirmed viral load <400 c/mL who had not met any non-responder criterion. Non-responders were PAR who never achieved confirmed HIV RNA <400 c/mL, prematurely discontinued study or study medication for any reason, had confirmed rebound to at least 400 c/mL, or had an unconfirmed HIV RNA of at least 400 c/mL at the last visit.
Time Frame: Week 24
Population: ITT-E Population. The primary analysis method was time to loss of virologic response (TLOVR) for the proportion of participants HIV-1 RNA <400 copies/mL at Week 24.
Measure: Number; unit: percentage of participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
percentage of participants | 88.4 | 86.6

5. Secondary Outcome: Percentage of Participants (PAR) Who Achieved Plasma HIV-1 RNA <400 c/mL at the Week 48 Visit: TLOVR Analysis
Description: The percentage of PAR with HIV-1 RNA virus <400 c/mL determined from blood samples drawn at Week 48 was tabulated by treatment arm with stratification by initial antiretroviral treatment. Per TLOVR algorithm, responders were PAR with confirmed viral load <400 c/mL who had not met any non-responder criterion. Non-responders were PAR who never achieved confirmed HIV RNA <400 c/mL, prematurely discontinued study or study medication for any reason, had confirmed rebound to at least 400 c/mL, or had an unconfirmed HIV RNA of at least 400 c/mL at the last visit.
Time Frame: Week 48
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
Percentage of participants | 81 | 84

6. Secondary Outcome: Percentage of Participants (PAR) Who Achieved Plasma HIV-1 RNA <400 c/mL at the Week 24 Visit: Observed, MD=F, and SNAPSHOT Analyses
Description: The percentage of PAR with HIV-1 RNA virus <400 c/mL determined from blood samples drawn at Week 24 was tabulated by treatment arm with stratification by initial antiretroviral treatment using specific analysis methods.
Time Frame: Week 24
Population: ITT-E Population. Analysis methods: (1) Observed: all observed data; (2) MD=F: PAR with missing data/data collected after study medication discontinuation (DC) were failures; (3) SNAPSHOT: PAR with missing data at Week 24/data collected after study medication DC/viral load >=400 c/mL were failures.
Measure: Number; unit: percentage of participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
percentage of participants
  Observed, n=181, 89 | 98.9 | 98.9
  M/D=F, n=199, 97 | 88.9 | 88.7
  SNAPSHOT, n=199, 97 | 89.4 | 89.7

7. Secondary Outcome: Percentage of Participants (PAR) Who Achieved Plasma HIV-1 RNA <400 c/mL at the Week 48 Visit: Observed, MD=F, and SNAPSHOT Analyses
Description: The percentage of PAR with HIV-1 RNA virus <400 c/mL determined from blood samples drawn at Week 48 was tabulated by treatment arm with stratification by initial antiretroviral treatment using specific analysis methods.
Time Frame: Week 48
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
Percentage of participants
  Observed, n=169, 82 | 96 | 100
  M/D=F, n=199, 97 | 81 | 82
  SNAPSHOT, n=199, 97 | 82 | 85

8. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 24
Description: Change from Baseline was calculated as the Week 24 value minus the Baseline value. Blood was drawn to analyze for plasma HIV viral load.
Time Frame: Baseline and Week 24
Population: ITT-E Population. Observed Population. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 24 visit and had a viral load result obtained during that visit period.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 181 | 89
log10 copies/mL | 0.014 (0.271) | 0.008 (0.352)

9. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 48
Description: Change from Baseline was calculated as the Week 48 value minus the Baseline value. Blood was drawn to analyze for plasma HIV viral load.
Time Frame: Baseline and Week 48
Population: ITT-E Population. Observed Population. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 48 visit and had a viral load result obtained during that visit period.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 169 | 82
log10 copies/mL | 0.071 (0.448) | -0.018 (0.198)

10. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24
Description: Blood was drawn to analyze for CD4+ cell count. A CD4+ cell is a T lymphocyte that carries the CD4 antigen. Immunologic response was assessed by CD4+ counts. Change from Baseline was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline and Week 24
Population: ITT-E Population. Observed Population. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 24 visit and had a CD4+ cell count obtained during that visit period.
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter (mm^3)
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 181 | 89
cells per cubic millimeter (mm^3) | 47.7 (134.02) | 8.3 (122.40)

11. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Description: Blood was drawn to analyze for CD4+ cell count. A CD4+ cell is a T lymphocyte that carries the CD4 antigen. Immunologic response was assessed by CD4+ counts. Change from Baseline was calculated as the Week 48 value minus the Baseline value.
Time Frame: Baseline and Week 48
Population: ITT-E Population. Observed Population. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 48 visit and had a CD4+ cell count obtained during that visit period.
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter (mm^3)
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 169 | 83
cells per cubic millimeter (mm^3) | 95.8 (158.93) | 57.2 (139.84)

12. Secondary Outcome: Change From Baseline in Fasting Triglycerides, Total Cholesterol, High-density Lipoprotein (HDL) Cholesterol, and Low-density Lipoprotein (LDL) Cholesterol at Week 24
Description: Triglycerides, total cholesterol, HDL cholesterol, and LDL cholesterol levels were measured at Week 24. A Fasting blood sample was drawn to analyze for lipids. Change from Baseline was calculated as the Week 24 value minus the Baseline value for each parameter.
Time Frame: Baseline and Week 24
Population: Safety Population: all randomized participants, with the exception of those with documented evidence of not having consumed any Investigational Product. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 24 visit and had a measurement taken during that visit period.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 170 | 81
milligrams per deciliter (mg/dL)
  Triglycerides, n=170, 81 | -17.23 (62.29) | -4.35 (63.00)
  Total cholesterol, n=170, 81 | 4.49 (26.37) | 0.14 (26.24)
  HDL cholesterol, n=170, 81 | 4.50 (8.78) | -0.20 (8.73)
  LDL cholesterol (Calculation), n=166, 80 | 3.34 (22.48) | 0.94 (25.72)

13. Secondary Outcome: Change From Baseline in Cholesterol/HDL Ratio at Week 24
Description: A Fasting blood sample was drawn to analyze for lipids. Change from Baseline was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 170 | 81
ratio | -0.20 (0.57) | -0.01 (0.66)

14. Secondary Outcome: Change From Baseline in Fasting Triglycerides, Total Cholesterol, High-density Lipoprotein (HDL) Cholesterol, and Low-density Lipoprotein (LDL) Cholesterol at Week 48
Description: Triglycerides, total cholesterol, HDL cholesterol, and LDL cholesterol levels were measured or calculated at Week 48. A fasting blood sample was drawn to analyze for lipids. Change from Baseline was calculated as the Week 48 value minus the Baseline value for each parameter.
Time Frame: Baseline and Week 48
Population: Safety Population: all randomized participants, with the exception of those with documented evidence of not having consumed any Investigational Product. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 48 visit and had a measurement taken during that visit period.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 152 | 76
milligrams per deciliter (mg/dL)
  Triglycerides, n=152, 76 | -9.28 (65.39) | 7.71 (91.00)
  Total cholesterol, n=152, 76 | 7.62 (31.04) | 0.62 (29.90)
  HDL cholesterol, n=152, 76 | 3.11 (9.33) | 0.53 (9.58)
  LDL cholesterol (Calculation), n=148, 71 | 5.28 (26.35) | -0.62 (28.21)

15. Secondary Outcome: Change From Baseline in Cholesterol/HDL Ratio at Week 48
Description: A fasting blood sample was drawn to analyze for lipids. Change from Baseline was calculated as the Week 48 value minus the Baseline value for each parameter.
Time Frame: Baseline and Week 48
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 152 | 76
ratio | 0.00 (0.97) | 0.00 (0.69)

16. Secondary Outcome: Number of Participants Who Met the Protocol-defined Confirmed Viral Failure Criteria Through Week 24
Description: The number of participants that failed to remain virologically suppressed through 24 weeks on treatment was assessed. Viral failure is defined per protocol as confirmed HIV-1 RNA >=400 c/mL.
Time Frame: From Baseline to Week 24
Population: ITT-E Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
participants | 2 | 1

17. Secondary Outcome: Number of Participants Who Met the Protocol-defined Confirmed Viral Failure Criteria Through Week 48
Description: The number of participants that failed to remain virologically suppressed from baseline through 48 weeks on treatment was assessed. Viral failure is defined per protocol as confirmed HIV-1 RNA >=400 c/mL.
Time Frame: From Baseline to Week 48
Population: ITT-E Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
participants | 4 | 1

18. Secondary Outcome: Number of Participants Who Experienced Death and/or Disease Progression
Description: Death and clinical disease progression (as per CDC classification) were assessed from Baseline through Week 48. Disease progression is defined as progression from CDC Class A to B, Class A to C, or from Class B to C. AIDS CDC classifications are: Class A, Asymptomatic/lymphadenopathy/acute HIV; Class B, Symptomatic, not AIDS; Class C, AIDS indicator conditions. The CDC categorization of HIV/AIDS is based on the lowest documented CD4 cell count (Class A, >=500 cells per microliter [µl]; Class B, 200-499 cells/µl; Class C, <200 cells/µl) and on previously diagnosed HIV-related conditions.
Time Frame: From Baseline to Week 48
Population: ITT-E Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
participants | 0 | 0

19. Secondary Outcome: Number of Confirmed Virologic Failure (VF) Participants (PAR) With Treatment-emergent HIV Genotypic Resistance in Reverse Transcriptase and Protease From Baseline Through Week 24
Description: A blood sample was drawn for particiapants with confirmed VF >=400 c/mL. For each participant, the mutations found at the time of failure were compared with any mutations found in the blood sample at Baseline. New resistance-associated viral mutations defined by the International Acquired Immunodeficiency Syndrome Society-United States of America guidelines present at the time of failure were tabulated by drug class. NRTI, nucleoside reverse transcriptase inhibitor; NNRTI, non-nucleoside reverse transcriptase inhibitor; PI, protease inhibitor.
Time Frame: From Baseline to Week 24
Population: ITT-E Population. Only those participants who met the confirmed VF criteria and had a viral genotype obtained at the time of VF were assessed.
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 2 | 1
participants
  PAR with treatment-emergent mutations | 2 | 1
  PAR with NRTI mutations | 1 | 0
  PAR with NNRTI mutations | 1 | 0
  PAR with major PI mutations | 1 | 0
  PAR with minor PI mutations | 2 | 1

20. Secondary Outcome: Number of Confirmed Virologic Failure (VF) Participants (PAR) With Treatment-emergent HIV Genotypic Resistance in Reverse Transcriptase and Protease From Baseline Through Week 48
Description: as for outcome 19
Time Frame: From Baseline to Week 48
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 4 | 1
participants
  PAR with treatment-emergent mutations | 4 | 1
  PAR with NRTI mutations | 2 | 0
  PAR with major NNRTI mutations | 1 | 0
  PAR with major PI mutations | 2 | 0
  PAR with minor PI mutations | 4 | 1

21. Secondary Outcome: Number of Confirmed Virologic Failure Participants (PAR) From Baseline Through Week 24 With the Indicated Treatment-emergent Reductions in Susceptibility to Abacavir, Lamivudine, Tenofovir, Emtricitabine, Atazanavir, or Ritonavir
Description: A blood sample was drawn for participants failing to respond to therapy, and changes in drug susceptibility for HIV isolated from the participants for each drug used in the study were assessed. For each participant, the changes in drug susceptibility detected by phenotypic assay in virus from the sample collected at the time of failure was compared with drug susceptibility in the virus from the blood sample at Baseline.
Time Frame: From Baseline to Week 24
Population: ITT-E Population. Only those participants who met the confirmed VF criteria with viral phenotype obtained at the time of virologic failure were assessed.
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 2 | 1
participants
  HIV PAR with reduced abacavir susceptibility | 1 | 0
  HIV PAR with reduced lamivudine susceptibility | 1 | 0
  HIV PAR with reduced tenofovir susceptibility | 0 | 0
  HIV PAR with reduced emtricitabine susceptibility | 1 | 0
  HIV PAR with reduced atazanavir susceptibility | 1 | 0
  HIV PAR with reduced ritonavir susceptibility | 1 | 0

22. Secondary Outcome: Number of Confirmed Virologic Failure Participants (PAR) From Baseline Through Week 48 With the Indicated Treatment-emergent Reductions in Susceptibility to Abacavir, Lamivudine, Tenofovir, Emtricitabine, Atazanavir, or Ritonavir
Description: as for outcome 21
Time Frame: From Baseline to Week 48
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 4 | 1
participants
  HIV PAR with reduced abacavir susceptibility | 1 | 0
  HIV PAR with reduced lamivudine susceptibility | 2 | 0
  HIV PAR with reduced tenofovir susceptibility | 0 | 0
  HIV PAR with reduced emtricitabine susceptibility | 2 | 0
  HIV PAR with reduced atazanavir susceptibility | 2 | 0
  HIV PAR with reduced ritonavir susceptibility | 2 | 0

23. Secondary Outcome: Number of Participants With the Indicated Grade 2 to Grade 4 Adverse Events (AEs) Occurring at a Frequency of >=3% in Either Treatment Group
Description: The National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 is a descriptive terminology that can be utilized for AE reporting. A grading (severity) scale is provided for each AE. Grade refers to the severity of the adverse event (AE). The CTCAE v3.0 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1, mild AE; Grade 2, moderate AE; Grade 3, severe AE; Grade 4, life-threatening or disabling AE; Grade 5, death related to the AE.
Time Frame: From Baseline to Week 24
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
participants
  Upper respiratory tract infection | 7 | 6
  Diarrhoea | 5 | 3
  Bronchitis | 4 | 3
  Rash | 6 | 0
  Muscle strain | 2 | 3
  Muscle spasms | 1 | 3
  Sinusitis | 1 | 3

24. Secondary Outcome: Number of Participants With the Indicated Grade 2 to Grade 4 Adverse Events (AEs) Occurring at a Frequency of >=3% in Either Treatment Group
Description: as for outcome 23
Time Frame: From Baseline to Week 48
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Number analyzed (Participants) | 199 | 97
participants
  Any Event | 90 | 44
  Upper respiratory tract infection | 11 | 7
  Diarrhoea | 7 | 4
  Depression | 6 | 3
  Back pain | 4 | 3
  Bronchitis | 4 | 3
  Insomnia | 6 | 0
  Muscle strain | 3 | 3
  Rash | 6 | 0
  Sinusitis | 2 | 4
  Muscle spasms | 2 | 3

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs occurring between the date of Randomization up to Week 48 are presented in this summary.
Arm/Group | ABC/3TC + ATV | TDF/FTC + ATV/RTV
Serious Adverse Events (participants affected / at risk) | 21/199 | 6/97
Other Adverse Events (participants affected / at risk) | 92/199 | 31/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABC/3TC + ATV (N=199) | TDF/FTC + ATV/RTV (N=97)
Cellulitis (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 2 | 0
Staphyloccal abscess (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 2 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABC/3TC + ATV (N=199) | TDF/FTC + ATV/RTV (N=97)
Nausea (Gastrointestinal disorders) | 28 | 4
Upper respiratory tract infection (Infections and infestations) | 22 | 12
Headache (Nervous system disorders) | 19 | 5
Diarrhoea (Gastrointestinal disorders) | 15 | 4
Rash (Skin and subcutaneous tissue disorders) | 15 | 1
Bronchitis (Infections and infestations) | 11 | 7
Insomnia (Psychiatric disorders) | 12 | 3
Sinusitis (Infections and infestations) | 9 | 7
Fatigue (General disorders) | 14 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 5

LIMITATIONS AND CAVEATS:
This study consists of a 35-day Screening Period, a 48-week Treatment Period, and a Follow-up Period (contact ~2-4 weeks after the Week 48/Withdrawal Visit). Data from Week 24 (primary endpoint) and Week 48 (final data) are presented in this summary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.